CLINICAL TRIAL: NCT02715167
Title: Predictive Factors in Response to Inhaled Corticoids in Chronic Cough
Acronym: FeNOTX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FeNOTX
Record Dates: First submitted 2016-03-04; First posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Group Budesonide (Active Comparator): Inhaled corticoids
  Interventions: Drug: Budesonide novolizer
- Group Placebo (Placebo Comparator): Placebo by inhalation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide novolizer
  Arms: Group Budesonide
Drug: Placebo
  Arms: Group Placebo

SUMMARY:
The hypothesis is that a high fractional exhaled nitric oxide can predict the response to inhaled corticoids in chronic cough.

ELIGIBILITY:
Inclusion Criteria:

* chronic cough

Exclusion Criteria:

* active smoker
* treated by corticoids during the previous month
* use of angiotensin-converting-enzyme inhibitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Leicester cough questionnaire | 5 minutes